CLINICAL TRIAL: NCT04958473
Title: A Single-center, Non-randomized Controlled, Single-arm, Phase II Clinical Trial of Sintilimab in Combination With Axitinib in the Treatment of Advanced Renal Cell Carcinoma
Brief Title: A Study of Sintilimab in Combination With Axitinib in Advanced Renal Cell Cancer
Acronym: SAARCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAARCC
Record Dates: First submitted 2021-06-23; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — sintilimab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with advanced RCC (Experimental): Patients with a diagnosis of kidney cancer (renal cell carcinoma, advanced or metastatic, previously treated or untreated)
  Interventions: Drug: Sintilimab; Drug: Axitinib

INTERVENTIONS:
Drug: Sintilimab — PD-1 inhibitor，Sintilimab 200mg IV, every 3 weeks.
  Other Names: Tyvyt; IBI 308
Drug: Axitinib — Tyrosine kinase inhibitor，licensed for use in treatment of renal cell carcinoma. Oral treatment Axitinib given 5 mg PO BID.
  Other Names: Inlyta

SUMMARY:
In patients with recurrent or metastatic renal cell carcinoma, a preliminary evaluation of the safety and efficacy of sintilimab combined with axitinib in patients with advanced renal cell carcinoma was conducted.Progression-free survival (PFS), overall survival (OS), disease control rate (DCR) and disease remission rate (ORR) were evaluated.

DETAILED DESCRIPTION:
Patients with recurrent or metastatic renal cell carcinoma received axitinib tablets (5mg bid po) combined with sintilimab (200mg d1) on a 3-week (21-day) as a one-cycle regimen.6 months of continuous administration (i.e., 8 cycles of sintilimab) or until tumor progression or unacceptable toxicity or death or subject withdraws informed consent;If the drug has been discontinued or the tumor has progressed, and there are no intolerable side effects, the drug can be continued according to the judgment of the researchers and the will of the subjects. Drug safety was evaluated before each cycle.The first efficacy was evaluated after 2 cycles.The efficacy was then evaluated every 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent before performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up
* Diagnosis of locally advanced or metastatic RCC that is predominantly clear cell histology
* Must have measurable disease
* Subject has received no prior systemic therapy
* A woman is eligible to participate in the study if she is of Non-childbearing potential, has a negative serum pregnancy test within 7 days of the first dose of study treatment, not lactating, and agrees to use adequate contraception during the study until at least 120 days after the last dose of investigational product
* Eastern Cooperative Oncology Group performance status 0 or 1
* Adequate organ function as defined in the protocol
* Left ventricular ejection fraction >= lower limit of normal as assessed by echocardiogram or multigated acquisition scan

Exclusion Criteria:

* Subject has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents
* Subject is currently participating or has participated in a study of an investigational agent or using an investigational device within 30 days of the first dose of study treatment
* Subject is expected to require any other form of systemic or localized antineoplastic therapy while on study
* Subject is on any systemic steroid therapy, within one week before the planned date for first dose of study treatment. Subject is on any other form of immunosuppressive medication
* Unable to swallow and retain orally administered medication
* Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other -Gastrointestinal conditions with increased risk of perforation; history of abdominal fistula, GI perforation, or intra-abdominal abscess within 4 weeks before beginning study treatment
* Known history of HIV infection or a known history of or is positive for Hepatitis B or Hepatitis C
* Presence of active infection requiring systemic therapy
* Corrected QT interval duration prolongation
* History of any one or more of the following cardiac conditions within the past 6 months: Cardiac angioplasty or stenting; Myocardial infarction; Unstable angina; ----History of Class III or IV congestive heart failure according to New York Heart Association classification
* History of cerebrovascular accident within the past 6 months
* Poorly controlled hypertension
* History of untreated deep venous thrombosis
* Presence of any non-healing wound, fracture, or ulcer, or presence of symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures
* Has taken any prohibited medications that are listed in the protocol within 14 days of the first dose of study treatment. Subject has received or will receive a live vaccine within 30 days before the first administration of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 12 months
  To be assessed by RECIST 1.1

SECONDARY OUTCOMES:
Progression free survival (PFS) | From randomization up to 3 years.
  Progression Free Survival (PFS) is the time from randomization to date of first documentation of objective progression of disease assessed by BICR (by RECIST version 1.1) or death due to any cause.
Overall Survival (OS) | Every 3 months up to 3 years.
  OS is the time from date of randomization to date of death due to any cause.
Disease Control Rate (DCR) | Every 6 weeks up to 18 months from patient enrollment in the study, then every 12 weeks up to 3 years from randomization
  DC is defined as complete response (CR), partial response (PR), or stable disease (SD) according to the RECIST v.1.1 recorded from randomization until disease progression assessed by BICR or death due to any cause.
Incidence of treatment-related adverse events | Up to 3 years.
  To be assessed by CTCAE v4.03.

CONTACTS AND LOCATIONS:
Overall Officials: BIN HUO, MD, Principal Investigator — Tianjin Medical University Second Hospital; Haitao Wang, PhD, Study Director — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No